CLINICAL TRIAL: NCT02446509
Title: A Psychoeducation Intervention for Caregivers of Patients With Bipolar Disorder: A Feasibility Study
Brief Title: A Psychoeducation Intervention for Caregivers of Patients With Bipolar Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Rebecca Lynn Casarez, Associate Professor - Clinical, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-SN-13-0579
Record Dates: First submitted 2015-04-23; First posted 2015-05-18 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Bipolar Disorder Family Members

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive a 7-week group psychoeducation intervention. Caregivers will meet once a week for 90-minute sessions in a group setting. Dates and times of the group sessions will be arranged according to the convenience of the subjects. The major content will include the causes of bipolar disorder, signs and symptoms of bipolar disorder, the role of stress and life events, types of medications and what they do, self-management of the disorder, understanding the course of the disorder, genetic and biological predispositions, how the family can help, management of relapse.
  Interventions: Behavioral: Psychoeducation
- Wait List Control Group (Active Comparator): Subjects in the wait list control group will receive the same 7 psychoeducation sessions after the experimental group receives these sessions.
  Interventions: Behavioral: Psychoeducation - Delayed

INTERVENTIONS:
Behavioral: Psychoeducation — Caregivers will meet once a week for 90-minute sessions in a group setting. Dates and times of the group sessions will be arranged according to the convenience of the subjects. The major content will include the causes of bipolar disorder, signs and symptoms of bipolar disorder, the role of stress and life events, types of medications and what they do, self-management of the disorder, understanding the course of the disorder, genetic and biological predispositions, how the family can help, management of relapse.
  Arms: Experimental Group
Behavioral: Psychoeducation - Delayed — The wait list control group will receive the same intervention as the experimental group, but 7 weeks later.
  Arms: Wait List Control Group

SUMMARY:
Bipolar disorder is a debilitating chronic illness characterized by periods of elation and depression. Since deinstitutionalization of the mentally ill over 40 years ago, families have become major caregivers for patients with bipolar disorder . This illness imposes a substantial and chronic burden on family caregivers Despite their persistent stress and burden, these caregivers have been largely ignored. Interventions to help them have been very limited. One comprehensive intervention was developed and implemented by Miklowitz (2008) and has shown to be effective in reducing caregiver depression and improving health outcomes. However, this intervention and is highly complex, long, and was given on an individual basis, significantly raising the cost of the program. One core component of the Miklowitz (2008) intervention is psychoeducation, which provides the fundamental support and information needed to caregivers on an individual basis.

In this pilot study, the intervention group will receive 7 weekly psychoeducation sessions. After completion of these sessions in the intervention group, the wait list control group will receive the same weekly sessions. In this study, the investigators plan to test the feasibility and potential efficacy of this specific psychoeducation intervention implemented in a group setting. The investigators will also examine the effects of this psychosocial intervention on biological mechanisms (cortisol and inflammatory biomarkers) and health outcomes.

The specific aims are to:

1. Test the feasibility of implementing a 7-week group psychoeducation program for family caregivers of patients with bipolar disorder by assessing recruitment and retention rates, attendance, satisfaction with the program, and data and sample collection rate.
2. Explore the effect of the intervention on caregiver outcomes (depression, burden, health status, mental wellbeing, cortisol, interleukin (IL)-1 and IL-6 levels.

The intervention will be delivered by at the University of Texas Health Science Center at Houston Center of Excellence for Mood Disorders (CEMD) and at the University of Texas Health Science Center at Houston School of Nursing. Forty family caregivers of patients with bipolar disorder will be recruited into the study.

ELIGIBILITY:
Inclusion Criteria:

* primary family caregiver of a patient with Bipolar Disorder who is age 16 or older;
* live within a 70 mile radius of the Center for Excellence in Mood Disorders (in the Texas Medical Center)

Exclusion Criteria:

* unstable major medical illness;
* health condition that may impact biomarker levels, e.g. is taking corticosteroids or anti-inflammatory drugs;
* unable to read, write, or speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Change in Caregiver Burden as measured by the Burden Assessment Scale at 8 weeks | Baseline, 8 weeks
Change in Caregiver Burden as measured by the Burden Assessment Scale at 16 weeks | Baseline, 16 weeks

SECONDARY OUTCOMES:
Change in Caregiver Mental Well Being as measured by the Warwick-Edinburgh Mental Well-Being Scale at 8 weeks | Baseline, 8 weeks
Change in Caregiver Mental Well Being as measured by the Warwick-Edinburgh Mental Well-Being Scale at 16 weeks | Baseline, 16 weeks
Change in Caregiver Depression as measured by the Quick Inventory of Depressive Symptomatology Clinician-Rated at 8 weeks | Baseline, 8 weeks
Change in Caregiver Depression as measured by the Quick Inventory of Depressive Symptomatology Clinician-Rated at 16 weeks | Baseline, 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at Houston School of Nursing, Houston, Texas, United States